CLINICAL TRIAL: NCT06722183
Title: FUTURE Platform Trial - A Phase II Platform Trial of Futibatinib in Combination With (Chemo)Immunotherapy in Colorectal Cancer and Other Solid Tumor Entities
Brief Title: Futibatinib in Combination With (Chemo)Immunotherapy in Colorectal Cancer and Other Solid Tumor Entities
Acronym: FUTURE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Universitätsmedizin Mainz, I. Medizinische Klinik, Forschungslabor Prof. Möhler (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUTURE; 2024-517573-24-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer
Keywords: platform trial; colorectal cancer; futibatinib; phase II
MeSH Terms: conditions — Colorectal Neoplasms | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Futibatinib plus tislelizumab plus mFOLFOX (Experimental): Futibatinib 20 mg orally, once daily, continuously, plus tislelizumab (i.v., 200 mg) on day 1 and day 22 at each 6-week cycle and mFOLFOX (SOC chemotherapy)
  Interventions: Drug: Futibatinib orally administered; Drug: Tislelizumab (i.v. 200mg)

INTERVENTIONS:
Drug: Futibatinib orally administered — Futibatinib will be administered 20mg orally, once daily, continously
Drug: Tislelizumab (i.v. 200mg) — Tislelizumab (i.v. 200mg) will be administered on day 1 and day 22 of a 6-week cycle

SUMMARY:
The FUTURE trial is a prospective, multicentre, exploratory, open-label phase II platform trial. Its goal is to evaluate the efficacy, feasibility and safety of futibatinib combined with immunotherapeutic, targeted or chemotherapeutic agents in colorectal and other solid tumors and to additionally identify biomarkers that correlate with clinical outcome.

DETAILED DESCRIPTION:
For the FUTURE-001 cohort:

All enrolled patients will take mFOLFOX 85 mg/m2 oxalipla n, 200 mg/m2 calcium folinate, 400 mg/m2 5-ﬂuorouracil as bolus dose and 2400 mg/m2 5-ﬂuorouracil as 48 h-infusion as standard chemotherapy on day 1, 15 and 29 of a 6-week cycle. Additionally, tislelizumab (i.v., 200 mg) is applied on day 1 and day 22. Futibatinib will be taken orally, once daily, continously. All patients enrolled will receive the study treatment for up to 12 months or until disease progression, unacceptable toxicity or patient's request or investigator's decision, whatever occurs first.

The primary objective is to evaluate the efficacy (primary endpoint: Overall Response Rate ORR, complete response + partial response) of futibatinib plus tislelizumab and chemotherapy in 1st-linetreatment of patients with colorectal cancer. The secondary objective is to evaluate further efficacy (duration of response (DoR, Progression-free survival (PFS), overall survival (OS)) as well as to assess safety and impact on the patients quality of life. Additionally, a correlation analysis between selected molecular parameters and clinical data to identify molecular biomarkers predictive for clinical outcome will be performed.

33 patients will be enrolled in this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patient* provides signed informed consent.
2. Patient is ≥ 18 years at the time of given informed consent.
3. Patient has a histologically proven solid tumor:

   • Specific for FUTURE-001: Histological or cytological confirmation of colorectal adenocarcinoma that is unresectable and/or metastatic with known RAS-, BRAF and MSI- status.
4. Specific for FUTURE-001: Patient must agree to participation in the accompanying translational research program.
5. Specific for FUTURE-001: Patient did not receive previous therapy in palliative setting (1st line situation).
6. Patient has ECOG Performance status ≤ 1.
7. Patient has adequate blood count, liver-enzymes, and renal function:

   1. ANC > 1,500 cells/μL without the use of hematopoietic growth factors
   2. Platelet count ≥ 100 x 109/L (>100,000 per mm3)
   3. Hemoglobin ≥ 9 g/dL, transfusion allowed
   4. Serum total bilirubin ≤ 1.5x institutional upper normal limit (ULN) (or < 2 x ULN in case of liver involvement or Gilbert's disease)
   5. AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional ULN without existing liver metastases, or ≤ 5 x UNL in the presence of liver metastases; AP ≤ 5 x ULN
   6. Patients not receiving therapeutic anticoagulation must have an INR ≤ 1.5 ULN and aPTT ≤ 1.5 ULN. The use of full dose anticoagulants is allowed as long as the INR or PTT is within therapeutic limits (according to the medical standard in the institution) and the patient has been on a stable dose for anticoagulants for at least three weeks at the time of inclusion
   7. Serum Creatinine ≤ 1.5 x ULN and a calculated creatinine clearance rate ≥ 50 mL /min
8. Patient has serum calcium and phosphate levels within normal range.
9. Female patients of childbearing potential or male patients with female partners of childbearing potential must agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of <1% per year during the treatment period and in FUTURE-001 for at least 1 week after last dose of futibatinib, 6 months after the last dose of chemotherapy or 4 months after last dose of tislelizumab, whatever is later. Male patients should refrain from sperm donation/ cryopreservation throughout this period and male patients with a pregnant partner must agree to remain abstinent or to use a condom for the duration of the pregnancy. Female patients of child-bearing potential must have a negative pregnancy test within the last 7 days prior to the start of trial therapy.
10. Patient is willing and able to comply with the protocol (including contraceptive measures) for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

    * There is no data that indicates a specific gender distribution. Therefore, patients are included regardless of their gender.

Exclusion Criteria:

1. Specific for FUTURE-001: Patient has curative colorectal cancer.
2. Patient received previous FGFR-addressed therapy with an FGFR inhibitor.
3. Patient has known presence of tumors other than the entity investigated in the respective cohort (FUTURE-001: colorectal cancer) or a secondary tumor other than squamous or basal cell carcinomas of the skin or in situ carcinomas of the cervix which have been effectively treated. The sponsor decides to include patients who have received curative treatment and have been disease-free for at least 5 years
4. Patient has known untreated or symptomatic CNS or leptomeningeal metastases.
5. Patient has history and/or current evidence of any of the following disorders:

   1. Non-tumor related alteration of the calcium-phosphorus homeostasis that is considered clinically significant in the opinion of the investigator
   2. Ectopic mineralization/calcification, including but not limited to soft tissue, kidneys, intestine, or myocardia and lung, considered clinically significant in the opinion of the investigator
6. Patient receives simultaneous, ongoing systemic immunotherapy, chemotherapy, or hormone anti-cancer therapy or any other anti-cancer treatment not described in the trial protocol (excluding palliative radiotherapy only for symptom control).
7. Patient has a stage B cirrhosis according to Child-Pugh criteria (or worse) or cirrhosis (of any grade) with a history of hepatic encephalopathy or clinically significant ascites resulting from cirrhosis. Clinically significant ascites is defined as ascites resulting from cirrhosis requiring diuretics or paracentesis.
8. Patient has known allergic / hypersensitive reactions to at least one of the treatment components.
9. Patient shows a ≥ grade 2 neuropathy
10. Patient takes St. Johns Wort within 6 weeks prior to initiation of study treatment
11. Patient has evidence of or any ongoing ophthalmological disorders. including but not limited to, central serous retinopathy, macular/retinal degeneration, diabetic retinopathy, and previous retinal detachment
12. Patient has other serious illnesses or medical ailments within the last 12 months prior to the start of the study.
13. Patient has a known presence of an active, uncontrollable infection.
14. Patient has active disseminated intravascular coagulation.
15. Patient has any other serious concomitant or medical condition that, in the opinion of the investigator, presents a high risk of complications to the patient or reduces the likelihood of clinical effect.
16. Patient participated in another interventional clinical study within 28 days prior to study enrollment or participation in a clinical study at the same time as this study, unless it is an observational/ non-interventional study or during the follow-up period of an interventional study.
17. Patient received treatment with any of the following within the specified time frame prior to the first dose of study treatment:

    1. Major surgery within 4 weeks (surgical incision should be fully healed)
    2. Radiotherapy for extended field within 4 weeks or limited field radiotherapy within 2 weeks
    3. Any investigational drug within 4 weeks
18. Female patients, who are pregnant or breast feeding or planning to become pregnant within 6 months after the end of treatment. Female patients of childbearing potential must have a negative serum pregnancy test result within 7 days prior to initiation of study treatment
19. Specific for FUTURE-001: Patient received prior treatment with PD-(L)1 or CTLA-4 targeted treatment
20. Specific for FUTURE-001: Patient has any active autoimmune disease or has a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis , hyperthyroidism; patients with vitiligo; asthma that has been completely remitted in childhood and does not require any intervention in adulthood can be included; patients with asthma requiring medical intervention with bronchodilators cannot be included)
21. Specific for FUTURE-001: Patient has immune deficiency or receives systemic steroid hormone therapy (> 10mg/day prednisone or other equivalents), or other form of immunosuppressive therapy within 2 weeks prior treatment initiation
22. Specific for FUTURE-001: Patient has history of uncontrolled infection with human deficiency virus (HIV) or chronic infection with hepatitis B or C virus (HBV, HCV)
23. Specific for FUTURE-001: Patient has received a solid organ transplantation
24. Specific for FUTURE-001: Patient has history of interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-12-16 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) according to RECIST v1.1 | up to 27 months
  ORR, defined as rate of patient who achieved complete or partial response (CR+PR) according to RECIST v1.1 as best response

SECONDARY OUTCOMES:
Duration of Response (DoR) | up to 27 months
  (DoR), defined as time from response initiation (when either CR or PR is first determined) to date of progression or death to any cause
Progression-free survival (PFS) according to RECIST v1.1 | every 8 weeks until disease progression, up to 27 months
  defined as time from date of enrollment to date of progression acc. to RECIST v1.1 or death due to any cause
Overall Survival (OS) | up to 27 months
  time from date of enrollment date of death due to any cause
Safety | AEs will be reported from start of trial treatment until 30 days after the last dose of study treatment or until initiation of another anti-cancer therapy, whichever occurs first, up to 13 months
  assessment of safety of the treatment as determined by the incidence, nature, causality, frequency, timing and severity of adverse events using NCI CTCAE 5.0

OTHER OUTCOMES:
Identifcation of molecular biomarkers | 27 months
  to perform correlation analysis between selected molecular parameters and clinical data to identify molecular biomarkers predictive for clinical outcome

CONTACTS AND LOCATIONS:
Overall Officials: Salah Al-Batran, Prof. Dr., Study Director — Institut für Klinische Krebsforschung IKF GmbH; Thorsten O. Götze, Prof. Dr., Principal Investigator — Institute of Clinical Cancer Research, UCT - University Cancer Center Frankfurt Krankenhaus Nordwest; Markus Möhler, Prof. Dr., Principal Investigator — Johannes Gutenberg-University Clinic Mainz
Locations (10):
- Germany (10):
  - Klinikum St. Marien Amberg, Amberg
  - Charité Campus Virchow Klinikum (CVK), Berlin
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Kliniken Essen-Mitte, Essen
  - Krankenhaus Nordwest, Frankfurt am Main
  - Hope Hamburg, Hamburg
  - Universitätsmedizin Mainz, Mainz
  - Klinikum München rechts der Isar, München
  - MVZ für Hämatologie und Onkologie Ravensburg GmbH, Ravensburg
  - Leopoldina Krankenhaus Schweinfurt, Schweinfurt

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared